CLINICAL TRIAL: NCT04791982
Title: The Study Was Conducted as a Pre-test-post-test, Control Group and Quasi-experimental Intervention Research Design in Order to Evaluate the Effects of Education Applied to Family Members Who Provide Care for Patients With Colorectal Cancer on Their Healthy Lifestyle Behaviors and Reactions Towards Caregiving. The Study Population Consisted of 100 Caregiver Who Provide Primary Care to Patients With Colorectal Cancer.
Brief Title: The Effect of Education Provided to Family Members Caring for Colorectal Cancer Patients on Caregiving Reactions and Healthy Lifestyle Behaviors: A Prospective Quasi-experimental Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Nilay Bektaş Akpınar, Associate professor, Ankara University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NBAkpınar
Record Dates: First submitted 2021-02-21; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Evaluation of the Effects of Education Provided on Family Members Caring for Colorectal Cancer Patients
Keywords: Caregiver; Caregiving reactions; Colorectal cancer; Family member; Educational program
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Behavioral: Educational sessions
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Educational sessions — Firstly, the literature was scanned and a education booklet prepared after the opinions of 5 academic nurses, who are experts in the field of oncology, was used. The booklet was included colorectal cancer treatment, symptoms that may develop due to chemotherapy and information on their control, psychosocial support of caregiving family members. Interviews and educational sessions with family members who agreed to participate in the study were held in one-on-one and face-to-face meeting room. These interviews lasted approximately 45 to 60 minutes for each family member. In the interviews, a educational booklet containing information on nutrition, exercise, symptom management, physical aspects of care and disease-specific care was used to present information to caregivers. All of educational sessions were performed by the single researcher.
  Arms: Experimental group

SUMMARY:
The effect of education provided to family members caring for colorectal cancer patients on caregiving reactions and healthy lifestyle behaviors: A prospective quasi-experimental study

DETAILED DESCRIPTION:
The study was conducted as a pre-test-post-test, control group and quasi-experimental intervention research design in order to evaluate the effects of education applied to family members who provide care for patients with colorectal cancer on their healthy lifestyle behaviors and reactions towards caregiving. The study population consisted of 100 caregiver who provide primary care to patients with colorectal cancer. The study data were collected using the "Socio-Demographic Characteristics Data Collection Form", "Healthy Lifestyle Behaviors Scale II (HPLP-II)" and the "Caregiver Reaction Assessment (CRA)". The pre-test was applied to the experimental and control groups at the first interview. The preferred interview format was a booklet. Three times face to-face individual educational sessions were provided to the experimental group, accompanied by a education booklet. After the third educational session the post-test was applied to the caregivers in the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers who committed to providing care to their patients diagnosed with Stage II/III CRC and agreed to participate in the study, and who were suitable to respond to the forms in terms of cognitive and mental health were included in the study.

Exclusion Criteria:

* Caregivers whose patients had previously received chemotherapy for CRC or had colostomy in their patients and who had previously been education on the subject were excluded from the study

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
The effects of education provided to family members caring for colorectal cancer patients receiving chemotherapy on Healthy Lifestyle Behaviors Scale. | through study completion, an average of 1 year.
  The change in the scala scores of the Healthy Lifestyle Behaviors Scale after the three face-to-face educational sessions provided to the experimental group accompanied by a education booklet compared to the pre-educational period.
  The minimum and maxmimum values of the scala are 52-208 and higher scores mean a better.
The effects of education provided to family members caring for colorectal cancer patients receiving chemotherapy on Caregiver Reaction Assessment Scala. | through study completion, an average of 1 year.
  The change in the scala scores of the Caregiver Reaction Assessment after the three face-to-face educational sessions provided to the experimental group accompanied by a education booklet compared to the pre-educational period.
  The minimum and maxmimum values of the scala are 24-120 and higher scores mean a worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Graduate School of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided